CLINICAL TRIAL: NCT02129218
Title: A Pilot Study to Determine the Feasibility of a Low Glycemic Load Diet in Patients With Stage I-III Colon Cancer
Brief Title: Low Glycemic Load Diet in Patients With Stage I-III Colon Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE7213; NCI-2014-00831 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE7213 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-04-17; First posted 2014-05-02 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Stage I Colon Cancer; Stage II Colon Cancer; Stage III Colon Cancer; Stage I Rectal Cancer; Stage II Rectal Cancer; Stage III Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Low glycemic load with standard diet (Experimental): Patients follow a low glycemic load diet with a standard dietary intervention for 12 weeks.
  Interventions: Other: questionnaire administration; Behavioral: Standard Dietary Intervention; Behavioral: Low glycemic load
- Cohort 2: Low glycemic load with intensified diet (Experimental): Patients follow a low glycemic load diet with intensified dietary intervention for 12 weeks.
  Interventions: Other: questionnaire administration; Other: laboratory biomarker analysis; Behavioral: Intensified Dietary Intervention; Behavioral: Low glycemic load
- Cohort 3: Medium glycemic load with standard diet (Active Comparator): Patients follow a medium glycemic load diet with standard dietary intervention for 12 weeks.
  Interventions: Other: questionnaire administration; Other: laboratory biomarker analysis; Behavioral: Standard Dietary Intervention; Behavioral: Medium Glycemic Load
- Cohort 4: Medium glycemic load with intensified diet (Active Comparator): Patients follow a medium glycemic load diet with intensified dietary intervention for 12 weeks.
  Interventions: Other: questionnaire administration; Other: laboratory biomarker analysis; Behavioral: Intensified Dietary Intervention; Behavioral: Medium Glycemic Load

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies including three day food record, twenty-four hour dietary recall, and a food acceptability questionnaire.
Other: laboratory biomarker analysis — Correlative studies
  Arms: Cohort 2: Low glycemic load with intensified diet; Cohort 3: Medium glycemic load with standard diet; Cohort 4: Medium glycemic load with intensified diet
Behavioral: Standard Dietary Intervention — Participants will be contacted by a nutritionist, in person every 2 weeks with phone contact on the alternating weeks. At the initial visit, each participant will be given verbal and written patient education materials, including low glycemic load diet recipes, meal plans, food preparation, and grocery shopping information. Individual instruction will be tailored to their baseline dietary preferences (e.g. vegan, allergies, etc).
  Arms: Cohort 1: Low glycemic load with standard diet; Cohort 3: Medium glycemic load with standard diet
Behavioral: Intensified Dietary Intervention — Patients will be contacted weekly, in person, by a nutritionist . Participants will take part in a cooking demonstration at the time of their initial visit. The demonstration will be hands-on and participants will be able to sample foods and recipes. In addition to grocery shopping information, participants will be accompanied by a nutritionist to their local grocery store to practice new shopping habits for their target dietary glycemic load. Each participant will also receive weekly random phone calls to assess his or her progress.
  Arms: Cohort 2: Low glycemic load with intensified diet; Cohort 4: Medium glycemic load with intensified diet
Behavioral: Low glycemic load
  Arms: Cohort 1: Low glycemic load with standard diet; Cohort 2: Low glycemic load with intensified diet
Behavioral: Medium Glycemic Load
  Arms: Cohort 3: Medium glycemic load with standard diet; Cohort 4: Medium glycemic load with intensified diet

SUMMARY:
This pilot clinical trial studies the feasibility of a low glycemic load diet in patients with stage I-III colon cancer. A low glycemic load diet includes foods that have low scores on the glycemic index. The glycemic index is a scale that measures how much a certain carbohydrate causes a person's blood sugar to rise. A low glycemic load diet may help decrease the chance of cancer coming back and improve the survival in patients with colon cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of following a low or medium glycemic load diet in patients with stage I-III (local-regional) colon cancer.

SECONDARY OBJECTIVES:

I. To determine patient-reported acceptability of diet. II. To determine nutritionist resources utilized. III. To evaluate the effect of lowering dietary glycemic load on body mass index (BMI), lipid metabolism and pro-oncogenic intermediaries of cellular metabolism.

OUTLINE: Patients are sequentially enrolled in 1 of 4 possible cohorts as needed based on the feasibility of the prior cohort.

COHORT 1: Patients follow a low glycemic load diet with standard dietary intervention (contact with nutritionist in person every 2 weeks with phone contact on the alternating weeks) for 12 weeks.

COHORT 2: Patients follow a low glycemic load diet with intensified dietary intervention (contact with nutritionist in person every week) for 12 weeks.

COHORT 3: Patients follow a medium glycemic load diet with standard dietary intervention for 12 weeks.

COHORT 4: Patients follow a medium glycemic load diet with intensified dietary intervention for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have stage I-III colon or rectal cancer and have undergone definitive therapy; definitive therapy may have included surgery alone, or surgery plus neoadjuvant and/or adjuvant therapy
* Patients must regularly consume a diet with a glycemic load > 150 as estimated through the 3 day food recall
* Patients must readily be available for a 3 month period and agree to participate in regular dietary adherence assessments (surveys and phone interviews)

Exclusion Criteria:

* Current participation in an intervention targeting diet or exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Individual patient compliance, defined by following assigned target glycemic load index >= 75% of the time between weeks 4 and 12 | Up to week 12
  This compliance rate will be determined through conducting a 24 hour telephone recall, every 2 weeks at random and calculating the glycemic load. For each dose cohort, the number and percentage of patients who are compliant will be summarized, with 90% confidence interval that accounts for the two-stage design.

SECONDARY OUTCOMES:
Food acceptability score | Up to 12 weeks
  Results of the acceptability survey will be tabulated and described (the questions use a 7 point likert scale), separately for each cohort.
Hours of nutritionist time per week | Up to 12 weeks
  The median number of hours will be calculated based on time spent with each patient, separately for each cohort.

OTHER OUTCOMES:
Change in serum levels of glycosylated hemoglobin | Baseline to up to 12 weeks
  Separately for each cohort, serum levels will be summarized descriptively and graphically across the follow-up period. Paired t-tests or Wilcoxon signed rank tests will be used to compare baseline vs. post-intervention levels of all biomarkers. Changes in biomarkers will be correlated with dietary glycemic index (GI) using Pearson or Spearman correlation coefficients, across the follow-up period.
Change in BMI | Baseline to up to 12 weeks
  Separately for each cohort, BMI levels will be summarized descriptively and graphically across the follow-up period.
Change in serum levels of markers of lipid metabolism | Baseline to up to 12 weeks
  Separately for each cohort, serum levels will be summarized descriptively and graphically across the follow-up period. Paired t-tests or Wilcoxon signed rank tests will be used to compare baseline vs. post-intervention levels of all biomarkers. Changes in biomarkers will be correlated with dietary GI using Pearson or Spearman correlation coefficients, across the follow-up period.
Change in serum levels of proteins affected by carbohydrate metabolism | Baseline to up to 12 weeks
  Separately for each cohort, serum levels will be summarized descriptively and graphically across the follow-up period. Paired t-tests or Wilcoxon signed rank tests will be used to compare baseline vs. post-intervention levels of all biomarkers. Changes in biomarkers will be correlated with dietary GI using Pearson or Spearman correlation coefficients, across the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Treasure, MD, Study Director — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio